CLINICAL TRIAL: NCT02080637
Title: Safety, Pharmacokinetics (PK) and Hemodynamic Effects of Ambrisentan in Single Ventricle Pediatric Patients
Brief Title: Ambrisentan in Single Ventricle
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kevin Hill (Other)
Responsible Party: Sponsor-Investigator, Kevin Hill, Assist Professor, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00050118
Record Dates: First submitted 2014-02-21; First posted 2014-03-06 (Estimated); Results first posted 2019-09-12 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-08

CONDITIONS: Hypoplastic Left Heart Syndrome; Hypoplastic Right-sided Heart Complex
Keywords: Single ventricle
MeSH Terms: conditions — Hypoplastic Left Heart Syndrome; Baetz-Greenwalt syndrome; Univentricular Heart | interventions — ambrisentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ambrisentan (Active Comparator): Oral ambrisentan 2.5 - 5 mg, single dose, once daily
  Interventions: Drug: Ambrisentan
- Placebo (Placebo Comparator): Oral placebo 2.5 - 5 mg, single dose, once daily
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ambrisentan — Once daily oral dosing
  Other Names: Leitaris
  Arms: Ambrisentan
Other: Placebo
  Arms: Placebo

SUMMARY:
Purpose: To evaluate the pharmacokinetics, bioavailability and hemodynamic efficacy of ambrisentan after Fontan surgical palliation of single ventricle heart defects.

Study activities and population group: Children undergoing Fontan surgical palliation for single ventricle defects will be eligible for the study. Up to 20 subjects will be enrolled (16 ambrisentan, 4 placebo) and will receive 3 days (3 doses) of ambrisentan starting on post-operative day #1 upon returning from the operating room. Ambrisentan plasma levels will be obtained at specified time points during treatment. Post-operative monitoring lines will be used to measure effects of ambrisentan on hemodynamics and pulmonary / systemic endothelial function.

DETAILED DESCRIPTION:
A. Purpose of the Study The purpose of the study is to evaluate the safety, pharmacokinetics (PK) and pharmacodynamics (PD) of ambrisentan in children with single ventricle heart defects that are undergoing Fontan (stage III) surgical palliation. This is a double blind, placebo controlled study. The primary objective of this Phase I/II study is to assess the plasma PK, safety and PD of oral ambrisentan in children with surgically palliated single ventricle heart defects. A secondary objective will be to assess whether ambrisentan improves post-operative outcomes including amount and duration of chest tube drainage and hospital length of stay.

B. Background and Significance Complex congenital heart defects associated with underdevelopment of a ventricle account for ~8% of congenital heart disease with a birth incidence of 4-8/10000 live births. These single ventricle lesions are associated with high morbidity and 5 year mortality rates that approach 50%. Staged surgical palliation directs returning venous blood flow directly into the lungs so that pulmonary blood flow occurs without the aid of a pumping chamber. The final stage of surgery (stage III - the Fontan procedure) incorporates inferior caval blood flow directly into the pulmonary arteries. Consequently pulmonary blood flow and cardiac output are directly related to pulmonary vascular resistance and ventricular function. The limitations of single ventricle surgical palliation often result in a prolonged post-operative course with pleural effusions a particular concern. There is also continued long term attrition. Elevated pulmonary vascular resistance and impaired systemic ventricular function are important risk factors for early and late failure of single ventricle palliation.

Ambrisentan is an endothelin receptor antagonist that improves pulmonary and possibly systemic endothelial function. Ambrisentan is approved for treatment of pulmonary arterial hypertension in adults and is used off-label for treatment of pulmonary hypertension in childen. Children with single ventricle heart defects demonstrate both pulmonary and systemic endothelial dysfunction and may benefit from treatment with this drug. However pharmacokinetics and hemodynamic efficacy of ambrisentan have not been studied in single ventricle patients. The most widely used alternative agent, sildenafil, was recently associated with increased mortality in children. There is now a Food and Drug Administration (FDA) safety warning against use of sildenafil in children. The investigators have previously demonstrated hemodynamic benefits with use of sildenafil in these patients but ambrisentan is a potentially safer agent. Therefore this study would fill an unmet need to guide dosing and evaluate efficacy of ambrisentan in this vulnerable population.

C. Design and Procedures

This is a single-center, randomized, blinded PK study of ambrisentan in children ages ≥ 24 months and ≤120 months with single ventricle anatomy. There will be up to 20 subjects enrolled; 16 will receive ambrisentan and 4 will receive placebo. A small placebo control group is warranted to ensure that any treatment effect is not a result of post-operative improvement. Patients will be enrolled at the time of their routinely scheduled Fontan surgery.

Initial Dose: Oral ambrisentan 2.5 - 5 mg, single dose, once daily (nasogastric and gastrostomy tube administration will be considered only when a nasogastric or gastrostomy tube is already in place as part of routine post-operative care).Subjects will be randomized by Investigational Drug Services (IDS) to placebo (n=4) or oral ambrisentan (n=16) using permuted blocks. Subjects will receive either an oral suspension (2.5 or 5mg) or a 5mg tablet depending on their ability to swallow a tablet. To begin to ensure safety, the initial 5 subjects enrolled in the study (at least 4 active drug) will receive a dose of 2.5mg in a liquid suspension prepared by IDS. After enrollment of these subjects the investigators will perform a preliminary PK/safety analysis and evaluate ambrisentan exposure. If the drug is well tolerated (no grade III or greater adverse events) and exposure is less than the target exposure of 500-800ng/mL, then the investigators may increase the dose to 5mg/dL provided via tablet in those able to take a tablet or suspension for all others. If drug exposure is less than 100ng/mL then the investigators will enroll additional study subjects to ensure that at least 16 study subjects achieve adequate drug exposure. If drug exposure is in the target range then the investigators will continue to enroll study subjects to receive the 2.5mg suspension.

The total study duration is expected to be approximately 24 months for enrollment of up to 20 subjects. Study participants will remain in the study until 1 month after discharge following stage III surgery intervention or for 6 months - whichever is shorter. The subjects will receive routine care before, during and immediately after surgery and after hospital discharge. The investigators will record all in-hospital adverse events and tabulate by organ system. One month after the last study drug administration (dose #3), the investigators will contact patients by phone or evaluate in person if they remain hospitalized.

Plasma PK will be evaluated using a limited sampling scheme. A preliminary safety and PK analysis will be performed after 5 subjects are enrolled. Ambrisentan PK will be evaluated and dosing may be adjusted to achieve levels consistent with those reported in the adult and pediatric literature.

D. Study Interventions:

Baseline/Pre-Dose Assessment

After the parent or legally authorized representative has signed the Internal Review Board (IRB) - approved informed consent form, and after it has been determined that the patient satisfies all inclusion and exclusion criteria, the following evaluations will be performed and recorded in the case report form (CRF):

1. Baseline demographics, medical history and medical baseline conditions.
2. Physical examination.
3. Preoperative laboratory assessment (obtained as part of usual clinical care for pre-operative assessment:

   1. Hematology: hematocrit, hemoglobin, white blood cell count with differential, platelet count.
   2. Serum chemistry: creatinine, blood urea nitrogen, sodium, potassium, calcium.
   3. Liver function tests: aspartate transaminase (AST), alanine transaminase (ALT), alkaline phosphatase, total bilirubin, conjugated bilirubin, serum albumin.

Study Procedures

1. Record the start and stop time of ambrisentan administration and all concomitant drugs.
2. Hemodynamic evaluation performed prior to initiation of study drug and at 0-1,1-6,18-30 and 40-60hrs after administration of the first ambrisentan dose (blood samples will be collected only if central monitoring lines remain or if they can be timed with a routine lab collection)

   1. Record Fontan, common atrial, and systemic arterial pressures from existing central lines that are placed as part of routine post-operative care.
   2. Collect study labs (coincident with scheduled PK levels - see below):

   i. plasma samples for biomarkers (endothelin 1 [ET1], brain natriuretic peptide [BNP]).

   c. Record oxygen saturation from routinely collected arterial and venous blood gases.

   d. Perform study echocardiogram at baseline and at one time point in the following 72hours at least 2 hours after ambrisentan administration.
3. PK blood samples (500 µL, up to 7 per patient) and pressure measurements will be obtained at baseline and at 1-2, 3-4, 5-6, 8-12, 12-16, 24, and 48-84 hours post-initial drug administration.
4. Adverse events will be collected during and for 1 month after the last study drug administration. Results will be tabulated by organ system.
5. Physical examination will be performed within 24 hours after administration of study drug and once daily during study enrollment.
6. Record all AEs and SAEs.
7. Record all concomitant medication administered 24 hours after administration of study drug.
8. Up to 4 scavenge samples will be obtained from the clinical laboratory from samples collected in the 24 hours following ambrisentan administration. Scavenged samples are left over heparinized plasma samples from these children that are collected from the clinical laboratory prior to discarding.

PK Sampling A limited PK sampling scheme will be employed such that no more than 3500 μl (7 samples, 500 μl per sample) of blood is obtained.

Hospitalization Procedures

1. Any of the following clinical laboratories performed as standard of care during the study will be recorded. The investigators will use the laboratory values closest to study dose if there have been multiple tests.

   1. Hematology: hematocrit, hemoglobin, white blood cell count with differential, platelet count
   2. Serum chemistry: creatinine, blood urea nitrogen, sodium, potassium, calcium
   3. Liver function tests: aspartate transaminase (AST), alanine transaminase (ALT), alkaline phosphatase, total bilirubin, conjugated bilirubin
2. Physical examination will be performed daily during the post-operative hospitalization.
3. Record all Adverse Events (AEs) for 24 hours after the last dose of study drug
4. Record all Serious Adverse Events (SAEs) for 1 month after the last dose of study drug
5. Record duration of mechanical ventilation
6. Record hospital length of stay
7. Record intensive care unit length of stay
8. Record duration and volume of chest tube drainage

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 24 months; ≤120 months.
2. History of congenital heart disease with severe hypoplasia of a right or left ventricle.
3. Undergoing Fontan surgery as part of standard clinical care.
4. Availability and willingness of the parent/legally authorized representative to provide written informed consent and, as appropriate, assent from the child.

Exclusion Criteria:

1. History of serious adverse event related to ambrisentan administration.
2. History of ambrisentan exposure within 48 hours of the study.
3. Presence of pulmonary venous obstruction.
4. Treatment with cyclosporin.
5. Any of the following - as determined by the attending physician

   * Significant hemodynamic instability
   * Sepsis.
   * Need for ECMO support.
6. Renal failure defined as serum creatinine > 2 times higher than the upper limit of normal.
7. Liver dysfunction defined as alanine aminotransferase or aspartate aminotransferase > 3 times higher than the upper limit of normal.
8. Thrombocytopenia defined as a platelet count < 50 000 cells/µL.
9. Leukopenia defined as white blood cells < 2500 cells/µL.
10. Anemia defined as hemoglobin < 8mg/dL.
11. Atrial hypertension (mean LA pressure > 12mm Hg).

Ages: 24 Months to 120 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2015-07; Primary Completion 2017-07-20 (Actual); Study Completion 2017-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Hill, MD, Principal Investigator — Duke University
Locations (1):
- Duke Universtiy Hospital, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Oral placebo 2.5 - 5 mg, single dose, once daily
  Placebo
Period: Overall Study
Arm/Group | Ambrisentan | Placebo
Started | 13 | 3
Completed | 13 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ambrisentan | Placebo | Total
Number analyzed (Participants) | 13 | 3 | 16
Age, Continuous [Mean (Standard Deviation); unit: months] | 35 (6.7) | 48 (20.5) | 37.4 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 7
  Male | 7 | 2 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 12 | 2 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 10 | 1 | 11
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 3 | 16

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve for Ambrisentan Plasma Concentration
Description: Plasma samples collected at 0-1,1-6,18-30 and 40-60 hours after administration of the first ambrisentan dose.
Time Frame: 0-1,1-6,18-30 and 40-60 hours
Population: Five participants did not have all samples collected. Outcome measure not applicable to the Placebo group.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Ambrisentan
Number analyzed (Participants) | 8
ng*hr/mL | 7871.46 (36.96)

2. Primary Outcome: Change in Pulmonary Vascular Resistance Index
Description: Hemodynamic data, including Fontan pressures, common atrial pressures and saturations, will be collected at the specified timepoints. Pressures and saturations will be measured from existing monitoring lines. Standard Fick calculations will be used to calculate pulmonary vascular resistance (calculated as trans-pulmonary gradient [Fontan pressure - atrial pressure] / pulmonary blood flow [Qp]) and reported in Wood Units x m^2.
Time Frame: baseline to 2 hours post ambrisentan administration
Population: One participant in the Ambrisentan group had central line removed early; Fontan pressures could not be measured.
Measure: Mean (Standard Deviation); unit: WU*m^2
Arm/Group | Ambrisentan | Placebo
Number analyzed (Participants) | 12 | 3
WU*m^2 | -0.5 (0.5) | -0.2 (0.5)
Statistical Analysis 1: Comparison: Ambrisentan; Baseline versus 2 hours post-ambrisentan; Test type: Other; p = 0.01, Paired t-test; Mean Difference (Final Values) = -0.5, Standard Deviation 0.5

3. Secondary Outcome: Amount of Chest Tube Drainage Post Fontan Operation
Description: Total chest tube drainage in mL in first 96hrs after Fontan
Time Frame: 0-96 hours post Fontan
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Ambrisentan | Placebo
Number analyzed (Participants) | 13 | 3
milliliters | 1325 (531) | 1356 (622)
Statistical Analysis 1: Comparison: Ambrisentan vs Placebo; Test type: Other; p = 0.94, Regression, Linear; Slope = -27, 95% CI 2-sided [-775 to 723]

4. Secondary Outcome: Duration of Chest Tube Drainage Post Fontan Operation
Description: Chest tube duration will be calculated as the number of days from placement to removal.
Time Frame: measured for the duration of the post-operative hospitalization or for 30 days, whichever is shorter
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Ambrisentan | Placebo
Number analyzed (Participants) | 13 | 3
days | 6.54 (3.9) | 5.33 (1.5)
Statistical Analysis 1: Comparison: Ambrisentan vs Placebo; Test type: Other; p = 0.61, Regression, Linear; Slope = 1.2, 95% CI 2-sided [-3.9 to 6.3]

ADVERSE EVENTS:
Time Frame: During hospitalization and for 30 days after administration of the last dose
Arm/Group | Ambrisentan | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/3
Other Adverse Events (participants affected / at risk) | 8/13 | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ambrisentan (N=13) | Placebo (N=3)
Electrolyte abnormalities (Metabolism and nutrition disorders) | 8 | 2
Anemia (Blood and lymphatic system disorders) | 2 | 0
Prolonged pleural effusion or chylothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Hypertension requiring treatment (Cardiac disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-21): https://cdn.clinicaltrials.gov/large-docs/37/NCT02080637/Prot_SAP_000.pdf